CLINICAL TRIAL: NCT05730894
Title: Predictors of Mortality in Patients With VA-Extracorporeal Membrane Oxygenation. A Retrospective Data Review.
Brief Title: Predictors of Mortality in Patients With VA-Extracorporeal Membrane Oxygenation.
Acronym: ECMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MRC-01-22-574
Record Dates: First submitted 2022-12-05; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-11

CONDITIONS: Morality; VA-ECMO
Keywords: mortality; VA-ECMO; outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Venoarterial extracorporeal membrane oxygenation (VA-ECMO) support is a lifesaving tool used to treat cardiogenic shock, acute heart failure, or extracorporeal cardiopulmonary resuscitation(CPR). However, its use is associated with significant complications, including mortality. We aim to conduct a retrospective observational study of all patients at Heart Hospital who required VA-ECMO support due to cardiogenic shock during 1/06/2016 and 1/06/2022 to report the incidence of in-hospital mortality among patients who required VA-ECMO along with the predictors of mortality. Data will be collected to identify baseline characteristics and outcomes including clinical variables predictive of poor outcomes.

DETAILED DESCRIPTION:
Extracorporeal membrane oxygenation (ECMO) is an advanced life support modality for critically ill patients with refractory cardiac or respiratory failure. It is a temporary support for cardiorespiratory failure, bridging time for recovery or permanent assist. Besides, ECMO could be used in a variety of clinical presentations, such as severe traumas, extracorporeal-assisted rewarming (ECAR) of accidental deep hypothermia, and can be used as a bridge to lung or heart transplant.

Cardiogenic shock can be a fatal condition with poor prognosis. Conventional treatments for cardiogenic shock include vasopressor agents guided by invasive monitoring, and intraaortic balloon pump support. There has been growing interest in the use of veno-arterial extracorporeal membrane oxygenation (VA-ECMO) as a salvage therapy for patients in cardiogenic shock refractory to conventional treatments. However, there is a low rate of survival to weaning or bridging therapy among patients with cardiogenic shock requiring ECMO (42-56%). Moreover, VA-ECMO use is associated with complications, including bleeding, renal failure. Thus, the benefits of this potentially life-saving support is still subject to discussion, especially for VA-ECMO use in the setting of cardiogenic shock as the evidence is scarce. Therefore, it important to identify the patients' related factors that may be associated with poor outcomes using real-world data. We will conduct a retrospective observational study of all patients at Heart Hospital who required VA-ECMO support due to cardiogenic shock during 1/06/2016 and 1/06/2022 with the aim of quantifying the incidence of in-hospital mortality among patients who required VA-ECMO in the setting of cardiogenic shock along with determining the predictors of mortality.

ELIGIBILITY:
Inclusion Criteria:

* Adults with the age of ≥ 18 years
* Requiring VA-ECMO or VAV-ECMO support

Exclusion Criteria:

* Requiring VV-ECMO support

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Requirement of VA-ECMO support
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-02-28 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
mortality | 6 months
  mortality in patients who had VA-ECMO

SECONDARY OUTCOMES:
bacterial pathogens responsible for infection-related mortality in VA-ECMO | 1 month
  infection

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad medical corporation, Doha, DA, Qatar